CLINICAL TRIAL: NCT05268341
Title: Neuroimaging Reveals Treatment-related Changes in DLD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Karla Washington, Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01DC019337 (NIH)
Record Dates: First submitted 2022-02-10; First posted 2022-03-07 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Developmental Language Disorder
MeSH Terms: conditions — Language Development Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): computer assisted intervention targeting expressive grammar for preschoolers with DLD
  Interventions: Behavioral: My Sentence Builder
- No treatment (No Intervention): business as usual classroom (educational) services

INTERVENTIONS:
Behavioral: My Sentence Builder — computer-assisted treatment program for expressive grammar
  Arms: Treatment

SUMMARY:
Children with developmental language disorders (DLD, aka specific language impairment), a prevalent pediatric disorder, experience hallmark grammar deficits with life-long impacts on educational and occupational outcomes. While effective and early interventions can mitigate the impact of DLD, not enough is known about the neural basis of DLD in young children, yet is needed to inform the design of more individualized interventions. This project uses neuroimaging, along with behavioral methods, with the goal of better understanding the memory-language mechanisms that underlie grammar learning and impairment, while also considering their association to treatment-related changes in preschoolers with DLD.

DETAILED DESCRIPTION:
Although the impact of developmental language disorder (DLD), a prevalent preschool disorder, can be mitigated through evidence-based and early interventions, little is known about the neural basis of DLD, especially in young children, yet is useful in the design of efficacious treatments. While much of the evidence has been furnished by studies examining domain-specific processes (language network), domain-general processes relating memory and language also offer valuable testing ground and present the opportunity to advance the current knowledge base. The Procedural circuit Deficit Hypothesis (PDH) posits that grammar deficits are explained by an impairment of procedural memory (rule learning, "knowing how"). This impairment is associated with structural abnormalities in connections between frontal brain regions and basal ganglia, with corresponding underactivation and reduced functional connectivity. However, the declarative memory system (semantic, "knowing what"), supported by cortical and subcortical regions in the temporal lobes, including hippocampus, is spared, acting as a compensatory mechanism to offset grammar deficits.

This proposed research will use neuroimaging (functional MRI and diffusion imaging) to describe the neural basis (functional and structural connectivity) of grammar learning and treatment-related change by way of the PDH. The investigators will gather critical data regarding grammar learning in preschoolers with DLD before, after, and following a break in intervention (computer-assisted treatment: DLD treatment; "business as usual": DLD no treatment) as part of a randomized controlled trial. The investigators will also include typically developing (TD) peers to inform development vs disorder. Our central hypothesis is that treatment designed to improve grammar learning will normalize the procedural learning network in association with increases in language function and that the degree of improvement may be associated with the underlying neurobiology of baseline grammar deficits.

Building on a robust history of recruitment and treatment of preschoolers with DLD, the investigators will enroll 184 preschoolers, 100 with DLD (n=50 treatment; n=50 no treatment controls) and 84 TD. Aim 1 will establish the relationship between functional and structural connectivity for preschoolers with DLD and their TD peers between regions in the procedural learning and declarative networks. In Aim 2, the investigators will establish the neurobiological basis of treatment-related changes in DLD only. The investigators examine potential changes in functional and structural connectivity between regions of the procedural learning and declarative memory networks, and investigate whether treatment-related changes occur into the typical range (DLD and TD). To meet our scientific goals, the investigators pair behavioral tools (traditional grammar tools) with neuroimaging to describe co-occurring behavioral performance underlying learning and outcome. This research will contribute novel insights into mechanisms underlying learning and impairment to help advance the evidence-based management of DLD.

ELIGIBILITY:
Inclusion Criteria:

* ages 48-71 months
* average nonverbal intelligence quotient (IQ)
* enrolled in participating center
* typically developing (receptive and expressive language, social, articulation, other)
* DLD for expressive grammar
* typical oral motor function
* typical social/pragmatics skills
* average hearing thresholds
* monolingual and native Standard English speakers
* does not have any uncorrected vision challenges

Exclusion Criteria:

* receiving co-occurring speech-language or other intervention for communication
* not MRI safe
* special education placement of child based on ability or behavior

Ages: 48 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 184 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Functional connectivity data (time 1) from typical and DLD preschoolers | Time 1 (pre)
  Aim 1 (all TD and DLD preschoolers)- Primary: Pre/Time 1 data for functional connectivity (assessed using fMRI from the Sentence Completion Expressive Language Task- Preschool (SCELT-P)) between Regions of Interest (ROI) in the procedural learning network and in the declarative memory network
Functional connectivity data DLD preschoolers only to assess changes with treatment | Pre-to-post (up to 14 weeks), post-to-followup (at 27 to 28 weeks)
  Primary: Pre-to-post changes and maintenance of changes post-to-followup in functional connectivity (assessed using fMRI from the SCELT-P) between ROI within the procedural learning network and within the declarative memory network.
Functional connectivity data for typically developing and DLD preschoolers to assess changes in development | pre-to-follow-up (up to 28 weeks)
  Changes in development (pre-to-followup) in functional connectivity (assessed using fMRI from the SCELT-P) between ROI within the procedural learning and declarative memory networks.

SECONDARY OUTCOMES:
Structural connectivity data for typically developing and DLD preschoolers | Pre/Time 1 (up to 3-weeks)
  Main Secondary: structural connectivity (assessed using diffusion imaging) between anatomically-selected ROI in the procedural learning and declarative memory networks
Structural connectivity data for DLD preschoolers only to assess changes with treatment | pre-to-post (up to 14-weeks) and post-to-follow-up (at 27 to 28 weeks)
  Main Secondary Pre-to-post changes and maintenance of changes post-to-followup in structural connectivity (assessed using diffusion imaging) between anatomically-selected ROI in the procedural learning network and declarative memory network
Structural connectivity data for typically developing and DLD preschoolers to assess development and disorder over time. | pre-to-followup (up to 28-weeks)
  Main Secondary: Changes in development (pre-to-followup) in structural connectivity (assessed using diffusion imaging) between anatomically-selected ROI in the procedural learning network and in the declarative memory network
Percent correct on a grammar task for typically developing and DLD preschoolers to assess development and disorder. | Pre/Time 1 (up to 3-weeks)
  Additional secondary outcomes raw score on the PI-designed 45-item grammar probe (%correct for each of the three target forms, 15-forms per target). Scores are combine to get a total score on the task
Raw score on the SPELT-3 for typically developing and DLD preschoolers to assess development | Pre/Time 1 (up to 3-weeks)
  Additional secondary outcomes raw score a standard grammar test (SPELT-3)
Raw score on the DSS for typically developing and DLD preschoolers to assess development | Pre/Time 1 (up to 3-weeks)
  Additional secondary outcomes raw score a standard play based task (DSS) to assess development and disorder
Percent correct on a grammar screener for DLD preschoolers only to identify treatment targets | Pre/Time 1 (up to 3-weeks)
  Additional secondary outcomes: raw change score on the PI-designed grammar probe
Percent correct on a grammar task for DLD preschoolers only | Pre-to-post (up to 14 weeks), post-to-followup (at 27 to 28 weeks)
  Additional secondary outcomes raw score on the PI-designed 45-item grammar probe (%correct for each of the three target forms, 15-forms per target). Scores are combine to get a total score on the task.
Raw score on the SPELT-3 for DLD preschoolers only to assess change with treatment | Pre-to-post (up to 14 weeks), post-to-followup (at 27 to 28 weeks)
  Additional secondary outcomes raw score a standard grammar test (SPELT-3)
Raw score on the DSS for DLD preschoolers only to assess change with treatment | Pre-to-post (up to 14 weeks), post-to-followup (at 27 to 28 weeks)
  Additional secondary outcomes raw score a standard play based task (DSS) to assess changes with treatment
Percent correct on a grammar task for typically developing and DLD preschoolers to assess development and disorder. | pre-to-followup (up to 28-weeks)
  Additional secondary outcomes raw score on the PI-designed 45-item grammar probe (%correct for each of the three target forms, 15-forms per target). Scores are combine to get a total score on the task
Raw score on the SPELT-3 for typically developing and DLD preschoolers to assess development | pre-to-followup (up to 28-weeks)
  Additional secondary outcomes raw score a standard grammar test (SPELT-3)
Raw score on the DSS for typically developing and DLD preschoolers to assess development | pre-to-followup (up to 28-weeks)
  Additional secondary outcomes raw score a standard play based task (DSS) to assess development and disorder

CONTACTS AND LOCATIONS:
Overall Officials: Karla N Washington, PhD, Principal Investigator — University of Cincinnati
Locations (6):
- United States (6):
  - New Horizon Childcare, Cincinati, Ohio
  - Empower Learn Create INC, Cincinnati, Ohio
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - CWFF CHild Development Center, Cincinnati, Ohio
  - Wesley Education Center for Children and Families, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No